CLINICAL TRIAL: NCT06124040
Title: Sexual Function, Coping and Dyadic Coping in Cervical Cancer Patients: a Comparison Between Surgery and Radiotherapy Plus Chemotherapy
Brief Title: Sexual Function, Coping and Dyadic Coping in Patients With Cervical Cancer
Acronym: SUCCEEDER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6044
Record Dates: First submitted 2023-10-24; First posted 2023-11-09 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-10

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radio-chemotherapy: Cervical cancer patients undergoing radio-chemotherapy.
  Interventions: Behavioral: psychological assessment evaluation
- Surgery: Cervical cancer patients undergoing surgery.
  Interventions: Behavioral: psychological assessment evaluation

INTERVENTIONS:
Behavioral: psychological assessment evaluation — A prospective data collection will be performed with self-administered psychological measures, with the aim to compare two different groups of patients with cervical cancer neo diagnosis, candidates for non conservative surgery or radio-chemotherapy treatment, based on FIGO Gynecologic Oncology Committee Guidelines.
  Test will be repeated at Time 0 (firs access in radiotherapy Day Hospital, or first access in hospital ward for surgery), and Time 1 (after 6 months).

SUMMARY:
The studies currently available in the literature about sexual function and coping in cervical cancer are poor and heterogeneous, and their results are often conflicting; therefore, no definitive recommendations can be formulated. Furthermore, it is unclear whether the dysfunction is attributable to surgical sequelae, radiotherapy, chemotherapy, or psychological aspects related to cancer. Moreover, a baseline evaluation about sexual function and coping if often lacking.

Aim of this protocol is to perform a prospective longitudinal study to compare surgical vs. radio-chemotherapy cervical cancer patients, with the following objectives:

* To assess sexual function, coping, emotional distress, and quality of life of patients with cervical cancer undergoing surgery vs radiotherapy plus chemotherapy.
* To evaluate changes on the previous variables over 6 months.

The results obtained will be utilized for:

* planning precocious psycho-educational interventions aimed at promoting psychological and couple well-being in cervical cancer patients since diagnosis
* develop tools and educational programs for more appropriate communication about intimacy between healthcare professionals and patients.

DETAILED DESCRIPTION:
Many recent reviews focused on QoL and the sexual function of patients with cervical cancer and have only evaluated the sexual dysfunctions of patients undergoing chemo-radiotherapy plus interventional radiotherapy.

The studies currently available in the literature are poor and heterogeneous, and their results are often conflicting; therefore, no definitive recommendations can be formulated. Furthermore, it is unclear whether the dysfunction is attributable to surgical sequelae, radiotherapy, chemotherapy, or psychological aspects related to cancer. In fact, psychological factors caused by the cancer diagnosismay also negatively influence sexual functioning independently of the type of treatment or stage of cancer.

Common psychological issues included poor body image, decreased sense of femininity, anxiety about sexual interactions, and pain.

Consequently, related social issues may emerge, for example, the ability to maintain a sexual relationship, communication difficulties, and adverse effects on intimate relationships.

Women with cervical cancer have thus independently significant issues related to sexual functioning as a result of their disease and/or its treatment. The most important classification for cervical cancer is FIGO (International Federation Gynecology and Obstetrics) updated in 2021. Treatments for cervical cancer are different depending on this classification. Although early-stage cervical cancers have different prognosis and treatments with respect to invasive cervical cancers (surgery vs chemoradiation plus interventional radiotherapy), both types can have a major impact on patients' sexual function and coping, also dyadic coping since diagnosis.

For this reason, we decided to perform a prospective longitudinal study to compare surgical vs. radio-chemotherapy cervical cancer patients, with the following objectives:

Primary objectives: to assess sexual function and coping Secondary objective: to evaluate emotional distress; dyadic coping; anxiety and depression; QoL of patients with cervical cancer; association between coping and possible dissociative symptoms; changes on the previous variables over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age ≥ 18 years
* Patients undergoing non-conservative surgery or radiotherapy plus chemotherapy
* Patients able to understand and sign informed consent

Exclusion Criteria:

* Patients' age > 65 years
* Patients with inability to express informed consent
* Patients denying informed consent
* Patients with psychopathological disturbances preexisting to the cancer diagnosis
* Patients affected by severe language deficits

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cervical cancer neo diagnosis, pertaining to the Gynecologic Oncology and Radiotherapy Oncology Units of Fondazione Policlinico Universitario A. Gemelli IRCCS, candidates for surgery or radio-chemotherapy treatment, based on FIGO Gynecologic Oncology Committee Guidelines.
  Based on the evidence in literature and the historical of our Institution (throughout the year 2022: 81 radiotherapy plus chemotherapy, 64 surgery), assuming a slightly lower mean difference in psychological tests scores between the two groups due to the recent improvement in irradiation techniques since the previous publication, we calculated the final sample size is 154 patients, 88 undergoing radiotherapy plus chemotherapy and 66 undergoing surgery.
Sampling Method: Probability Sample
Enrollment: 154 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Assess sexual function in cervical cancer patients | 6 months. Time 0: the day of the beginning of the treatment (surgery or radio-chemotherapy), and Time 1: 6 months from the first assessment.
  Primary outcome is to assess sexual function of cervical cancer patients undergoing surgery vs patients undergoing radiotherapy plus chemotherapy.
  This dimension will be assessed by "Female Sexual Function Index" (FSFI), a survey measuring the sexual functioning of women in six different domains: desire, arousal, lubrication, orgasm, satisfaction and pain. The index only measures sexual function in these domains over the previous 30 days.
  The FSFI can be used as a screening tool and as a potential diagnostic aid. A total cut-off score ≤ 26.55 has been proposed for the diagnosis of female sexual dysfunction, so any woman scoring below 26.55 should be considered at risk for sexual dysfunction.
Assess individual coping strategies in cervical cancer patients | 6 months. Time 0: the day of the beginning of the treatment (surgery or radio-chemotherapy), and Time 1: 6 months from the first assessment.
  Assessment of individual coping strategies will be done in both groups by The Mini-Mental Adjustment to Cancer (Mini-MAC), a 29-item instrument that evaluates cognitive and behavioral responses to cancer. The factors of the Mini-MAC are: Fighting Spirit, Hopelessness, Anxious Preoccupation, Fatalism, and Cognitive Avoidance. Each item is rated on a 4-point scale that ranges from "definitely does not apply to me" to "definitely applies to me".
  Each statement is rated on a scale from 1 (definitely not) to 4 (definitely yes), and the available scores for each of the four coping strategies range from 7 to 28 points.
  The higher the score, the greater the coping/behavior style in the patient's fight against cancer.

SECONDARY OUTCOMES:
Evaluate dyadic coping in cervical cancer patients | 6 months. Time 0: the day of the beginning of the treatment (surgery or radio-chemotherapy), and Time 1: 6 months from the first assessment.
  Dyadic Adjustment Scale (DAS) will be adopted to assess the quality of romantic relationships in both patient and her partner, if any.
  This tool evaluates the adaptability, quality, and representation that each partner has with regard to an intimate relationship. It is a self-reporting questionnaire consisting of 32 items, divided into four subscales: dyadic satisfaction, dyadic cohesive, dyadic and affective consent.
  For this test there is not a real clinical cut-off, the higher the score the greater the cohesion within the couple. Minimum and maximum scores depend on the subscales:
  * Suscale CONSENT ON IMPORTANT ISSUES: minimum score 0, maximum 4
  * Subscale SATISFACTION WITH THE STATUS OF THE RELATIONSHIP: minimum score 0, maximum 5
  * Subscale DOING TOGETHER: minimum score 0, maximum 4
  * Subscale SATISFACTION FOR AFFECTIVE AND SEXUAL LIFE: minimum score 0, maximum 5
Evaluate emotional Distress in cervical cancer patients | 6 months. Time 0: the day of the beginning of the treatment (surgery or radio-chemotherapy), and Time 1: 6 months from the first assessment.
  Both groups will be administred by Distress Thermometer (DT), to evaluate emotional distress.
  Clinical cut-off are considered as follow:
  DT: > or = 4 (scoring equal or higher than 4 means high emotional distress).
Evaluate Anxiety and Depression in cervical cancer patients | 6 months. Time 0: the day of the beginning of the treatment (surgery or radio-chemotherapy), and Time 1: 6 months from the first assessment.
  Both groups will be administred by Hospital Anxiety and Depression Scale (HADS), to evaluate anxiety and depression.
  Clinical cut-off are considered as follow:
  HADS: 8-10 (a score lower than 8 means physiological levels of anxiety and depression; scores between 8 and 10 means the presence of anxiety and depression; scoring higher than 10 means high levels of anxiety and depression).
Evaluate the presence of any dissociative symtoms in cervical cancer patients | 6 months. Time 0: the day of the beginning of the treatment (surgery or radio-chemotherapy), and Time 1: 6 months from the first assessment.
  The Dissociative Experience Scale (DES-II) measures a wide variety of dissociation types, including both problematic experiences and normal experiences (e.g., daydreaming). It is a screening tool for dissociative disorders, especially dissociative identity disorder and dissociative disorder not otherwise specified.
  It is a 28-item questionnaire answered on a percentage scale ranging from 0% to 100%.
  The total score can be between 0 and 100, and is obtained by dividing the global result by the number of items.
  Scores higher than 30 indicate high levels of dissociation and are frequently reported in psychiatric patients with dissociative symptoms, while scores higher than 40 are related to post-traumatic stress disorder.
  Dissociation occupies an important position in the genesis of emotional manifestations in patients affected by cancer.
  In cancer, dissociative or post-traumatic symptoms can be related to coping strategies of anxious preoccupation and cognitive avoidance.
Evaluate quality of life dimensions in cervical cancer patients | 6 months. Time 0: the day of the beginning of the treatment (surgery or radio-chemotherapy), and Time 1: 6 months from the first assessment.
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Cervical Module (EORTC QLQ - CX24) is a Quality of Life questionnaire, designed to assess disease-specific and treatment-specific aspects of QoL in patients with cervical cancer.
  The QLQ-CX24 consists of 3 multi-item scales and 5 single-item scales which analyzed 3 dimensions: Symptom Experience; Body Image; Sexual/Vaginal Functioning.
  All subscales have a minimum score of 0 (no symptoms) and a maximum score of 4 (high presence of symptoms). In general, high scores indicate dysfunctional or pathological characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Agostino Gemelli IRCCS, Roma, RM, Italy